CLINICAL TRIAL: NCT03554408
Title: A Phase 1, Dose Escalation, First-in-human Study of the Safety and Pharmacokinetics of the Subcutaneous and Intravenous Administration of 10-1074-LS Alone and in Combination With 3BNC117-LS in HIV-infected and HIV-uninfected Individuals
Brief Title: First-in-human Study of 10-1074-LS Alone and in Combination With 3BNC117-LS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YCO-0971
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: 10-1074-LS; 3BNC117-LS; First in Human; Dose Escalation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Antibodies, Monoclonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Groups 1A, 1B, 4A, and 4B are double-blinded; All other arms are open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Group 1A (Experimental): HIV-uninfected individuals will be administered one 1 mL (approximately 150 mg) subcutaneous injection of 10-1074-LS or placebo (formulation buffer), in a 3:1 ratio.
  Interventions: Drug: 10-1074-LS
- Group 1B (Experimental): HIV-uninfected individuals will be administered one 2 mL (approximately 300 mg) subcutaneous injection of 10-1074-LS or placebo (formulation buffer), in a 3:1 ratio.
  Interventions: Drug: 10-1074-LS
- Group 2A (Experimental): HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS dosed at 3 mg/kg.
  Interventions: Drug: 10-1074-LS
- Group 2B (Experimental): HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS dosed at 10 mg/kg.
  Interventions: Drug: 10-1074-LS
- Group 2C (Experimental): HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS dosed at 30 mg/kg.
  Interventions: Drug: 10-1074-LS
- Group 3B (Experimental): HIV-infected individuals (on ART) will be administered one intravenous infusion of 10-1074-LS dosed at 10 mg/kg
  Interventions: Drug: 10-1074-LS
- Group 3C (Experimental): HIV-infected individuals (on ART) will be administered one intravenous infusion of 10-1074-LS dosed at 30 mg/kg.
  Interventions: Drug: 10-1074-LS
- Group 4A (Experimental): HIV-uninfected individuals will be administered one 2 mL (approximately 150 mg of each mAb) subcutaneous injection of 10-1074-LS admixed with 3BNC117-LS or placebo (formulation buffer), in a 3:1 ratio.
  Interventions: Drug: 10-1074-LS; Drug: 3BNC117-LS
- Group 4B (Experimental): HIV-uninfected individuals will be administered two 2 mL (approximately 300 mg of each mAb) subcutaneous injections of 10-1074-LS admixed with 3BNC117-LS or placebo (formulation buffer), in a 3:1 ratio.
  Interventions: Drug: 10-1074-LS; Drug: 3BNC117-LS
- Group 5 (Experimental): HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS and one intravenous infusion of 3BNC117-LS, each dosed at 30 mg/kg.
  Interventions: Drug: 10-1074-LS; Drug: 3BNC117-LS
- Group 6 (Experimental): HIV-infected individuals (on ART) will be administered one intravenous infusion of 10-1074-LS and one intravenous infusion of 3BNC117-LS, each dosed at 30 mg/kg.
  Interventions: Drug: 10-1074-LS; Drug: 3BNC117-LS
- Group 7 (Experimental): HIV-uninfected individuals will be administered three subcutaneous injections of 10-1074-LS (100 mg) admixed with 3BNC117-LS (200 mg) (2 mL) at weeks 0, 12, and 24.
  Interventions: Drug: 10-1074-LS; Drug: 3BNC117-LS
- Group 8 (Experimental): HIV-infected individuals (on ART) will be administered three subcutaneous injections of 10-1074-LS (75 mg) admixed with 3BNC117-LS (225 mg) (2 mL) at weeks 0, 12, and 24.
  Interventions: Drug: 10-1074-LS; Drug: 3BNC117-LS
- Group 9 (Experimental): HIV-infected individuals (on ART) will be administered three subcutaneous injections of 10-1074-LS (60 mg) admixed with 3BNC117-LS (250 mg) (2 mL) at weeks 0, 12, and 24.
  Interventions: Drug: 10-1074-LS; Drug: 3BNC117-LS

INTERVENTIONS:
Drug: 10-1074-LS — Subcutaneous injection of 10-1074-LS
  Other Names: Monoclonal antibody
  Arms: Group 1A; Group 1B; Group 4A; Group 4B; Group 7; Group 8; Group 9
Drug: 10-1074-LS — Intravenous infusion of 10-1074-LS
  Other Names: Monoclonal antibody
  Arms: Group 2A; Group 2B; Group 2C; Group 3B; Group 3C; Group 5; Group 6
Drug: 3BNC117-LS — Subcutaneous injection of 3BNC117-LS
  Other Names: Monoclonal antibody
  Arms: Group 4A; Group 4B; Group 7; Group 8; Group 9
Drug: 3BNC117-LS — Intravenous infusion of 3BNC117-LS
  Other Names: Monoclonal antibody
  Arms: Group 5; Group 6

SUMMARY:
This first clinical study of 10-1074-LS will evaluate its safety, tolerability and pharmacokinetics profile when administered alone or in combination with 3BNC117-LS to HIV (human immunodeficiency virus) -infected and HIV-uninfected individuals.

DETAILED DESCRIPTION:
The proposed study is a Phase 1, dose escalation cohort study of 10-1074-LS alone or in combination with 3BNC117-LS, administered intravenously and subcutaneously in HIV uninfected and HIV-1 infected individuals.

Study participants will be administered a single intravenous infusion of 10-1074-LS at 3, 10 or 30 mg/kg, single infusions of the combination of 10-1074-LS and 3BNC117-LS, each dosed at 30 mg/kg, or subcutaneous injections of 10-1074-LS alone or in combination with 3BNC117-LS, and three subcutaneous injections of 10-1074-LS in combination with 3BNC117-LS at three dose ratios. The first four groups administered subcutaneous injections of the product(s) will be randomized, double-blinded, and placebo-controlled to assess potential differences in safety and tolerability of the antibody formulation versus the formulation buffer alone. In the dose ratio portion of the study, participants will be randomized into one of three groups, but the products will be administered in an open-label manner. Groups administered intravenous infusions will be enrolled in an open-label manner.

PART A

Group 1A (n=8) - HIV-uninfected individuals will be administered one 1 mL (approximately 150 mg) subcutaneous injection of 10-1074-LS or placebo (formulation buffer), in a 3:1 ratio.

Group 1B (n=8) - HIV-uninfected individuals will be administered one 2 mL (approximately 300 mg) subcutaneous injection of 10-1074-LS or placebo (formulation buffer), in a 3:1 ratio.

Group 2A (n=3) - HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS dosed at 3 mg/kg.

Group 2B (n=3) - HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS dosed at 10 mg/kg.

Group 2C (n=3) - HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS dosed at 30 mg/kg.

Group 3B (n=3) - HIV-infected individuals (on ART) will be administered one intravenous infusion of 10-1074-LS dosed at 10 mg/kg.

Group 3C (n=3) - HIV-infected individuals (on ART) will be administered one intravenous infusion of 10-1074-LS dosed at 30 mg/kg.

PART B

Part B will begin after the Safety Monitoring Committee (SMC) evaluates available safety data from Part A, as detailed below. The SMC will also review available safety data with 3BNC117-LS administered intravenously collected under protocol YCO-0946 prior to enrollment in Part B of this study. The SMC will also review subcutaneous dosing at approximately 150 mg (1 mL) and 300 mg (2 mL), collected under IND 131873 when available and prior to enrollment in Part B of this study.

Group 4A (n=8) - HIV-uninfected individuals will be administered one 2 mL (approximately 150 mg of each mAb) subcutaneous injection of 10-1074-LS admixed with 3BNC117-LS or placebo (formulation buffer), in a 3:1 ratio.

Group 4B (n=8) - HIV-uninfected individuals will be administered two 2 mL (approximately 300 mg of each mAb) subcutaneous injections of 10-1074-LS admixed with 3BNC117-LS or placebo (formulation buffer), in a 3:1 ratio.

Group 5 (n=5) - HIV-uninfected individuals will be administered one intravenous infusion of 10-1074-LS and one intravenous infusion of 3BNC117-LS, each dosed at 30 mg/kg.

Group 6 (n=5) - HIV-infected individuals (on ART) will be administered one intravenous infusion of 10-1074-LS and one intravenous infusion of 3BNC117-LS, each dosed at 30 mg/kg.

Group 7 (n=6) HIV-uninfected individuals will be administered three subcutaneous injections of 10-1074-LS (100 mg) admixed with 3BNC117-LS (200 mg) (2 mL).

Group 8 (n=6) HIV-uninfected individuals will be administered three subcutaneous injections of 10-1074-LS (75 mg) admixed with 3BNC117-LS (225 mg) (2 mL).

Group 9 (n=6) HIV-uninfected individuals will be administered three subcutaneous injections of 10-1074-LS (60 mg) admixed with 3BNC117-LS (240 mg) (2 mL).

Following mAb or placebo administration, study participants will return for safety assessments on days 1 and 3, and weeks 1, 2 and 4 following each dose, then bi-monthly or monthly until the end of study follow up.

All participants will be followed for 48 weeks after last mAb or placebo administration. Serum samples for PK measurements will be collected before and at the end each mAb or placebo administration and at multiple subsequent time points during study follow up.

Samples will also be collected for measurement of HIV-1 plasma RNA levels before 10-1074-LS and 3BNC117-LS infusions and at follow up visits according to protocol.

ELIGIBILITY:
Inclusion Criteria:

Groups 1A-1B, 2A-2C, 4A-4B, 5, 7, 8, 9 (HIV-uninfected):

* Males and females, age 18 to 65
* Amenable to HIV risk reduction counseling and agrees to maintain behavior consistent with low risk of HIV exposure.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use two effective methods of contraception (i.e.

condom with spermicide, diaphragm with spermicide, hormone-eluting IUD, hormone-based contraceptive with condom) from 10 days prior to and nine months after 10-1074-LS and/or 3BNC117-LS administration.

- Female study participants of reproductive potential are defined as pre-menopausal women who have not had a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy). Women are considered menopausal if they have not had a menses for at least 12 months and have a FSH of greater than 40 IU/L or if FSH testing is not available, they have had amenorrhea for 24 consecutive months.

Groups 3B-3C, 6 (HIV-infected):

* Males and females, age 18 to 65.
* Confirmed HIV-1 infection.
* HIV-infected individuals on ART with HIV-1 plasma RNA levels < 50 copies/mL.
* Current CD4+ T cell count > 300 cells/μl.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy or transmission of HIV, agrees to use two effective methods of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting IUD, hormone-based contraceptive with condom) from 10 days prior to and nine months after 10-1074-LS and/or 3BNC117-LS administration.

Exclusion Criteria:

Groups 1A-1B, 2A-2C, 4A-4B, 5, 7, 8, 9 (HIV-uninfected):

* Confirmed HIV-1 or HIV-2 infection.
* Weight > 110 kg (subcutaneous groups only: 1A-1B, 4A-4B).
* History of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases) that in the opinion of the investigator would preclude participation.
* Within the 12 months prior to enrollment, the participant has a history of sexually transmitted infection.
* Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
* Laboratory abnormalities in the parameters listed:
* Absolute neutrophil count ≤ 1,500 cells/μL;
* Hemoglobin ≤ 11 gm/dL if female; ≤ 12.5 gm/dL if male;
* Platelet count ≤ 125,000 cells/μL;
* ALT ≥ 1.25 x ULN;
* AST ≥ 1.25 x ULN;
* Alkaline phosphatase ≥ 1.5 x ULN;by the trial physician within the last 6 months.
* Pregnancy or lactation.
* Any vaccination within 14 days prior to mAb infusions.
* Receipt of any experimental HIV vaccine or monoclonal antibody therapy of any kind in the past.
* History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
* Individuals with known hypersensitivity to any constituent of the investigational products.
* Receipt of another investigational product currently or within the past 12 weeks, or expected concurrent participation in another study in which investigational products will be administered.

Groups 3B-3C, 6 (HIV-infected):

* Have a history of AIDS-defining illness within 3 years prior to enrollment.
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases), other than HIV infection, that in the opinion of the investigator would preclude participation.
* Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
* Laboratory abnormalities in the parameters listed below:
* Absolute neutrophil count ≤ 1,000 cells/μl;
* Hemoglobin ≤ 10 gm/dL;
* Platelet count ≤ 100,000 cells/μl;
* ALT ≥ 1.5 x ULN;
* AST ≥ 1.5 x ULN;
* Alkaline phosphatase ≥ 1.5 x ULN;
* Total bilirubin > 1 x ULN;
* eGFR < 60 mL/min/1.73m2.
* Pregnancy or lactation.
* Any vaccination within 14 days prior to MAb infusions.
* Receipt of any experimental HIV vaccine or monoclonal antibody therapy of any kind in the past.
* History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
* Individuals with known hypersensitivity to any constituent of the investigational products.
* Receipt of another investigational product currently or within the past 12 weeks, or expected concurrent participation in another study in which investigational products will be administered.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
The number of participants who experience adverse events within 2 weeks after 10-1074-LS intravenous infusions and subcutaneous injections. | 2 weeks
  Adverse events include signs, symptoms and laboratory abnormalities, in addition to local and systemic reactogenicity adverse events.
The number of participants who experience adverse events within 2 weeks after 10-1074-LS and 3BNC117-LS intravenous infusions and subcutaneous injections. | 2 weeks
  Adverse events include signs, symptoms and laboratory abnormalities, in addition to local and systemic reactogenicity adverse events.
Elimination half-life (t1/2) of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups. | 48-72 weeks
  Elimination half-life (t1/2) of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups.
The clearance (CL) of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups. | 48-72 weeks
  The clearance (CL) of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups.
The volume of distribution (Vz) of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups | 48-72 weeks
  The volume of distribution (Vz) of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups
Area under the curve of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups. | 48-72 weeks
  Area under the curve of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups.
Decay curve of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups. | 48-72 weeks
  Decay curve of 10-1074-LS, when administered alone and in combination with 3BNC117-LS in all study groups.

SECONDARY OUTCOMES:
Frequency of induced anti-10-1074-LS antibodies | 48-72 weeks
  Frequency of induced anti-10-1074-LS antibodies
Level of induced anti-10-1074-LS antibodies | 48-72 weeks
  Level of induced anti-10-1074-LS antibodies
Frequency of induced anti-3BNC117-LS antibodies | 48-72 weeks
  Frequency of induced anti-3BNC117-LS antibodies
Level of induced anti-3BNC117-LS antibodies | 48-72 weeks
  Level of induced anti-3BNC117-LS antibodies
The number of participants that experience who experience adverse events during the study follow up period after 10-1074-LS and/or 3BNC117-LS administration in all study groups. | 48-72 weeks
  Adverse events include signs, symptoms and laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valente PK, Wu Y, Cohen YZ, Caskey M, Meyers K. Behavioral and social science research to support development of educational materials for clinical trials of broadly neutralizing antibodies for HIV treatment and prevention. Clin Trials. 2021 Feb;18(1):17-27. doi: 10.1177/1740774520948042. Epub 2020 Aug 24. PMID 32838558